CLINICAL TRIAL: NCT05415995
Title: A Prospective, Multicenter, Randomized Controlled Trail Using Drug-coated Balloon to Treat Below The Knee Arterial Stenosis or Occlusion
Brief Title: A Trail of Drug-coated Balloon Treating Below The Knee Arterial Diseases
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Zylox Medical Device Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: V1.1/2021-12-25
Record Dates: First submitted 2022-06-06; First posted 2022-06-13 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2022-03

CONDITIONS: Peripheral Artery Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 101 Patients with Below The Knee Artery stenosis or occlusion in Experimental Group (Experimental): Patients in this group use Drug eluting Balloon (Zylox-tonbridge), this is the product to be test in this clinical trail. The drug we coated is paclitaxel.
  Interventions: Device: Drug eluting Balloon
- 101 Patients with Below The Knee Artery stenosis or occlusion in Controlled Group (Active Comparator): Patients in this group use Drug eluting Balloon(Acotec), this is a product that has got approved by NMPA in 2016.
  Interventions: Device: Drug eluting Balloon

INTERVENTIONS:
Device: Drug eluting Balloon — Drug eluting Balloon is a kind of the product that has been used for many years. By filling the micropores on the surface of the balloon with anti-proliferative drugs like immunosuppressive agents, the balloon is expanded and contacted with the lesion to rapidly release the drug to the local arterial wall.

SUMMARY:
This is a prospective, multicenter, randomized controlled trail using drug-coated balloon to treat below the knee arterial stenosis or occlusion.

DETAILED DESCRIPTION:
This trail is conducted in several centers all around China. 202 subjects with below the knee arterial stenosis or occlusion will be recruited and randomized, this trail compares the efficacy and safety of Drug-coated Balloon (Zylox-Tonbridge) with a similar balloon catheter producted by Acotec. The subjects will be followed up when discharged /in 30 days/ 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-85 years；
* ≥70% diameter stenosis or occlusion in the target below-the-knee lesion；
* Rutherford Category 3-6；
* Subjects are willing to sign informed consent；

Exclusion Criteria:

* Planned major limb amputation within 30 days after the procedure;
* In-stent stenosis in the target lesion;
* Severely calcified target lesions；
* Creatinine>2.5mg/dL;
* History of allergies to anesthetics, contrast agents；
* Subjects who have participated in any other drug or medical device clinical investigations and haven't reach the primary endpoint；
* Other circumstances judged by researchers that are not suitable for enrollment.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Rate of primary patency of the target lesion | 180 days
  Primary patency is defined as no target lesion occlusion, no clinical symptom driven target lesion revascularization and major limb amputation.

SECONDARY OUTCOMES:
Success rate of the device | Intraoperation
  Success rate of the device is defined as a situation that the balloon catheter reached the lesion site, dilated successfully without rupture, and was successfully withdrawn.
Success rate of the technique | Immediately after the intervention
  On the basis of device success,technique success rate is defined as restored blood flow in the lesion after the treatment, and the residual stenosis ≤30%.
Success rate of the operation | Within 7 days
  On the basis of technique success, operation success is defined as no adverse event happening.

OTHER OUTCOMES:
Change of Ankle-Branchial Index(ABI) | 180 days
  ABI is a simple measurement identifies unrecognized Peripheral Arterial Disease.
The rate of target lesion revascularization(TLR) | 30 days/ 180 days
  TLR is defined as revascularization of the target lesion with stenosis ≥70%.

CONTACTS AND LOCATIONS:
Overall Officials: Junmin Bao, Principal Investigator — Changhai Hospital
Locations (20):
- China (20):
  - The second hospital of Anhui Medical university, Hefei, Anhui
  - Zhongshan Hospital Xiamen University, Xiamen, Fujian
  - Hebei General Hospital, Shijiazhuang, Hebei
  - The First Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - HeNan Province People's Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital Of Zhengzhou University, Zhengzhou, Henan
  - The central hospital of Wuhan, Wuhan, Hubei
  - Nanjing Drum Tower Hospital, the affiliated hospital of Nanjing University medical school, Nanjing, Jiangsu
  - The First Affiliated Hospital Of Dalian Medical University, Dalian, Liaoning
  - General Hospital of Northern Theater Command, Shenyang, Liaoning
  - The affiliated Hospital of QingDao University, Qingdao, Shandong
  - Shanxi Bethune Hospital, Taiyuan, Shanxi
  - The affiliated hospital of southwest medical university, Luzhou, Sichuan
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - Affiliated HangZhou First People's Hospital, Zhejiang University School of medicine, Hangzhou, Zhejiang
  - Huamei hospital, University of Chinese academy of sciences, Ningbo, Zhejiang
  - China-Japan Friendship Hospital, Beijing
  - Peking University First Hospital, Beijing
  - Changhai Hospital, Shanghai
  - Shanghai Ninth People's Hostpital, Shanghai JiaoTong University School of Medicine, Shanghai